CLINICAL TRIAL: NCT00526071
Title: Open-label Extension Study to Evaluate the Long-term Safety, Tolerability and Pharmacodynamics of AT1001 in Patients With Fabry Disease
Brief Title: Open-label Long-term Safety Study of AT1001 (Migalastat Hydrochloride) in Participants With Fabry Disease Who Have Completed a Previous AT1001 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor (Amicus Therapeutics) terminated this study for logistical reasons.
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB-CL-205
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Fabry Disease
Keywords: Amicus Therapeutics; AT1001; Galafold; Migalastat; Substrate
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Migalastat (Experimental): Migalastat was administered orally, 150 mg QOD, 250 mg QD for 3 days, 4 days off per week for 2 months, or 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site. Participants received migalastat for up to 56 months.
  Interventions: Drug: migalastat HCl

INTERVENTIONS:
Drug: migalastat HCl
  Other Names: AT1001; Galafold; migalastat

SUMMARY:
Study to evaluate the long-term safety, tolerability, and pharmacodynamics (PD) of migalastat hydrochloride (HCl) (migalastat) in participants with Fabry disease

DETAILED DESCRIPTION:
This was a long-term open-label study of migalastat in participants with Fabry disease who were previously enrolled in a Phase 2 study of migalastat (FAB-CL-201 [NCT00214500], FAB-CL-202 [NCT00283959], FAB-CL-203 [NCT00283933], or FAB-CL-204 [NCT00304512]). Participants could enter this extension study immediately upon completion of participation in their previous study of migalastat, or at a later time point. Thus, some participants did not necessarily have continuous treatment with migalastat from the end of the original study to the time of enrollment into this extension study. Participants who enrolled before Protocol Amendment 2 received migalastat 150 milligrams (mg) orally once every other day (QOD). After the amendment, these participants entered a dose escalation period (DEP) at their next scheduled visit. During the DEP, participants received migalastat 250 mg (once daily [QD] for 3 days and 4 days off per week) for the first 2 months. If there were no safety concerns, the dose was then increased to 500 mg QD for 3 days and 4 days off per week). Participants received 500 mg (QD for 3 days and 4 days off per week) for up to 10 months, depending on the approval date of the protocol amendments at each site. An interim review of safety and PD data was performed after all enrolled participants had completed at least 4 months of treatment in the DEP. After the review, the dose and regimen of migalastat was returned to 150 mg QOD for all participants, except those who were on another dose as previously agreed by the investigator and medical monitor.

The sponsor (Amicus Therapeutics) discontinued Study FAB-CL-205 for logistical reasons and not due to either safety concerns or lack of efficacy. Participants who were ongoing in Study FAB-CL-205 at the time of discontinuation were offered participation in another open-label, long-term treatment study of migalastat (AT1001-041 [NCT01458119]). Participants who did not enroll in Study AT1001-041 were contacted by telephone or another suitable method approximately 1 month after the End of Study (EOS) visit to inquire about adverse events and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed another Phase 2 study of migalastat in Fabry Disease
* Women of childbearing potential must have had a negative result on their pregnancy test
* Male and female participants agreed to use a reliable method of contraception during study treatment and for 4 weeks after study treatment termination
* Were willing and able to provide written informed consent

Exclusion Criteria:

* Had not completed a Phase 2 study of migalastat in Fabry Disease
* Had a major protocol violation in the preceding migalastat trial and was discontinued
* Had undergone or was scheduled to undergo kidney transplantation or was currently on dialysis
* Had been treated with another investigational drug (except migalastat) within 30 days of study start
* Had been treated with Fabrazyme® (agalsidase beta), Replagal™ (agalsidase alfa), Glyset® (miglitol), or Zavesca® (miglustat) within 2 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2012-09-08 (Actual); Study Completion 2012-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (8):
- United States (3):
  - Decatur, Georgia
  - New York, New York
  - Dallas, Texas
- Parkville, Australia
- Porto Alegre, Brazil
- Garches, France
- United Kingdom (2):
  - London
  - Salford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open label, long-term extension study for participants who completed one of 4 preceding Phase 2 studies (FAB-CL-201 [NCT00214500], FAB-CL-202 [NCT00283959], FAB-CL-203 [NCT00283933], or FAB-CL-204 [NCT00304512]). Participants could enter this study directly upon completion of the previous study or at a later point.
Pre-assignment Details: This study included a dose escalation period (DEP), in which migalastat was administered at 250 milligrams (mg) for 2 months. If there were no safety concerns the dose was increased to 500 mg for up to 10 months, depending on the date of amendment approval. Before and after the DEP, all but 1 participant (post-DEP 300 mg instead) received 150 mg.
Groups:
- Migalastat: Participants received migalastat 150 mg given orally once every other day (QOD) before and after the DEP. During the DEP participants received 250 mg once daily (QD) for 3 days, 4 days off per week for 2 months then 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site. One participant received migalastat 300 mg (QD for 3 days and 4 days off per week) until the end of the study.
Period: Overall Study
Arm/Group | Migalastat
Started | 23
Safety Population (All participants who received at least 1 dose of study drug) | 23
Pharmacodynamic (PD) Population (Received study drug and had a baseline measurement and at least 1 postbaseline PD measure) | 23
Amenable Population; Men (Amenable mutations based on the clinical trial (CT) Human Embryonic Kidney (HEK) assay) | 11
Amenable Population; Women (Amenable mutations based on the CT-HEK assay) | 5
Non-amenable Population; Men (Those without mutant forms of α-Gal A responsive to migalastat treatment based on the CT-HEK assay) | 3
Non-amenable Population; Women (Those without mutant forms of α-Gal A responsive to migalastat treatment based on the CT-HEK assay) | 4
Completed | 17
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Response to Study Drug | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Migalastat: Participants received migalastat 150 mg given orally QOD before and after the DEP. During the DEP participants received 250 mg QD for 3 days, 4 days off per week for 2 months then 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site. One participant received migalastat 300 mg (QD for 3 days and 4 days off per week) until the end of the study.
Arm/Group | Migalastat
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) with start date on or after administration of study drug or pre-existing conditions that worsened on or after the start of the first study drug administration (on Day 1). A severe AE was defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced one or more severe TEAEs after dosing on Day 1 through End of Study (EOS) or follow-up (for participants who did not enroll in Study AT1001-041) are presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through EOS (up to 56 months) or follow-up (28 days after EOS)
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Migalastat
Number analyzed (Participants) | 23
Participants | 9

2. Secondary Outcome: Absolute Change From Baseline In α-Galactosidase A (α-Gal A) Activity In Leukocytes To Month 42
Description: The activity of the α-Gal A enzyme was measured in leukocyte lysate by a validated fluorometric assay method, using 4-methylumbelliferone as a reference. The activity values obtained were normalized to protein (measured using a colorimetric assay). Baseline was defined as the last non-missing pre-treatment value for each participant in his or her respective preceding migalastat Phase 2 study. A negative change from Baseline indicates that α-Gal A activity decreased. α-Gal A activity levels are presented for Baseline and Month 42.
Time Frame: Baseline, Month 42
Population: PD Population: all participants who received at least 1 dose of study drug and who had a baseline measurement and at least 1 postbaseline PD measure.
Measure: Mean (Standard Deviation); unit: nanomoles (nm)/hour (hr)/mg protein
Groups:
- Amenable Population; Men: Amenable participants were those with mutant forms of α-Gal A determined to be responsive to migalastat treatment based on the CT-HEK assay. Migalastat was administered orally, 150 mg QOD before and after the DEP. During the DEP participants received 250 mg QD for 3 days, 4 days off per week for 2 months then 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site. One participant received migalastat 300 mg (QD for 3 days and 4 days off per week) until the end of the study.
- Amenable Population; Women: Amenable participants were those with mutant forms of α-Gal A determined to be responsive to migalastat treatment based on the CT-HEK assay. Migalastat was administered orally, 150 mg QOD before and after the DEP. During the DEP participants received 250 mg QD for 3 days, 4 days off per week for 2 months then 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site.
- Non-amenable Population; Men; Non-amenable Population; Women: Non-amenable participants were those without mutant forms of α-Gal A as determined by the CT-HEK assay. Migalastat was administered orally, 150 mg QOD before and after the DEP. During the DEP participants received 250 mg QD for 3 days, 4 days off per week for 2 months then 500 mg QD for 3 days, 4 days off per week for up to 10 months, depending on the approval date of the protocol amendments at each site.
Arm/Group | Amenable Population; Men | Amenable Population; Women | Non-amenable Population; Men | Non-amenable Population; Women
Number analyzed (Participants) | 11 | 5 | 3 | 4
nanomoles (nm)/hour (hr)/mg protein
  Baseline | 2.08 (2.433) | 16.84 (7.955) | 0.09 (0.047) | 14.62 (8.944)
  Month 42: number analyzed (Participants) | 7 | 3 | 0 | 4
  Month 42 | 7.88 (8.691) | 18.31 (14.186) |  | 9.77 (5.071)

3. Secondary Outcome: Pharmacokinetics Of Migalastat As Assessed By Plasma Concentration
Description: The concentration of migalastat was evaluated in plasma following a dose of 250 mg and 500 mg. Blood samples were taken at trough (predose or Time 0; just prior to the third dose during a 3 day on, 4 days off dosing regimen) and at peak (3 hr postdose; after the third dose during a 3 day on, 4 days off dosing regimen) during the Day 1 (250 mg) and Month 2 (500 mg) visits. This outcome presents the lowest and highest concentrations of migalastat measured in any of the participants for predose and 3 hr postdose.
Time Frame: 0 (predose on Day 1; start of DEP), 3 hr (postdose at Month 2; during DEP])
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Number; unit: nanograms/milliliter
Arm/Group | Migalastat
Number analyzed (Participants) | 23
nanograms/milliliter
  Predose Lowest Concentration | 5.94
  Predose Highest Concentration | 313
  250 mg 3 hr Postdose Lowest Concentration | 908
  250 mg 3 hr Postdose Highest Concentration | 5250
  500 mg 3 hr Postdose Lowest Concentration | 113
  500 mg 3 hr Postdose Highest Concentration | 8500

ADVERSE EVENTS:
Time Frame: Day 1 after dosing through EOS (up to 56 months) or follow-up (28 days after EOS). Follow-up was not required for participants who enrolled in Study AT1001-041.
Arm/Group | Migalastat
Serious Adverse Events (participants affected / at risk) | 7/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=23)
Atrial Fibrillation (Cardiac disorders) | 2
Atrial Flutter (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Sensation of Foreign Body (General disorders) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Migalastat (N=23)
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 4
Cystitis (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Abdominal pain upper (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Influenza like illness (General disorders) | 2
Irritability (General disorders) | 2
Pain (General disorders) | 2
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 4
Paraesthesia (Nervous system disorders) | 3
Migraine (Nervous system disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Platelet count increased (Investigations) | 2
Weight increased (Investigations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Palpitations (Cardiac disorders) | 5
Sinus bradycardia (Cardiac disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Limb injury (Injury, poisoning and procedural complications) | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Insomnia (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Vision blurred (Eye disorders) | 3
Vitamin d deficiency (Metabolism and nutrition disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Fabry's disease (Congenital, familial and genetic disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can only publish the results from this trial provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review. If requested, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.